CLINICAL TRIAL: NCT02243163
Title: Effect of Yoga on Life Quality and Immunity in Breast Cancer Patients After Operation and or Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1020106
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Female Breast Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga exercise (Experimental): Subjects will receive regular 90-minutes yoga classes twice a week for 3 months.
  Interventions: Behavioral: Yoga exercise

INTERVENTIONS:
Behavioral: Yoga exercise — Subjects will receive regular 90-minutes yoga classes twice a week for 3 months.

SUMMARY:
The purpose of study is to investigate if yoga exercise improve life quality and immune status in breast cancer patients after complete treatment (including surgery and / or radiotherapy and / or chemotherapy)

DETAILED DESCRIPTION:
It is well-known that exercise promote immune regulation for better life quality. However, the mechanism for better immunity and life quality is not clear. We postulate that Ayurveda yoga might benefit breast cancer women with completion of operation and/or chemotherapy and radiotherapy. The benefits could be due to immune modulation, and improve health perception and life quality, and even potential decrease of cancer relapse.

The study patients will do yoga twice a week for 12 weeks. The study primary endpoints are 1) to improve personal health perception, 2) to improve life quality and 3) to enhance human immunity. The study secondary endpoint will follow up the immunity changes 3 months after the intervention.

We anticipate to reach the primary endpoints and to publish the primary results in one year, the secondary endpoint will complete in the second year.

ELIGIBILITY:
Inclusion Criteria:

* Able to attend yoga program weekly, and fill out inform consent.
* Patients with breast cancer after complete treatment for at least 3 months (including surgery and / or radiotherapy and/or chemotherapy).

Exclusion Criteria:

* male
* overweight
* unable to do yoga exercise.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Improve personal health and life quality | Change from baseline in personal health and life quality at 6 months.
  Health and life quality will assessed by modified fatigue inventory and EORTC QLQ-C30 (version 3) at three different times: (1)baseline data: before yoga exercise, (2)outcome data: at 6 and 12 weeks post-test.

SECONDARY OUTCOMES:
Immune modulation | Change from baseline in human immunity at 3 months.
  Lymphocytes will be extracted from peripheral blood for analyses of lymphocytes subpopulation (Th1/ Th2/ Treg/ Th17), polarization (T-bet/ Gata-3/ Foxp3/ RORrt) and its related cytokines (Th1: IL-12/ IFN-γ/ IL-27; Th2: IL-4/ IL-13/ IL-25; Th17: IL-17A/ IL-6/ IL-21; Treg: TGF/ IL-10. Saliva collection for analyses of cortisol and IL-6 at 3 different times: (1) baseline data: before yoga exercise, (2)outcome data: at 6 and 12 weeks post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hui Yeh, PhD, Study Chair — Chang Bing Show Chwan Memorial Hospital & Central Taiwan University of Science and Technology; Kuender D. Yang, PhD, Study Director — Chang Bing Show Chwan Memorial Hospital; Shin-Mae Wang, MD., Principal Investigator — Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan